CLINICAL TRIAL: NCT01230827
Title: A Multicenter, Double-Blind, Randomized-Withdrawal Trial of Subcutaneous Golimumab, a Humanized Anti-TNFa Antibody, in Subjects With Active Polyarticular Juvenile Idiopathic Arthritis (JIA) Despite Standard Therapy
Brief Title: A Study of the Safety and Efficacy of CNTO 148 (Golimumab) in Children With Juvenile Idiopathic Arthritis (JIA) and Multiple Joint Involvement Who Have Poor Response to Methotrexate (GO KIDS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial has failed to meet primary - and major secondary endpoints
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017089; CNTO148JIA3001 (Other: Janssen Research & Development, LLC); 2009-015019-42 (EudraCT Number); NCT01777399 (obsolete NCT alias)
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; golimumab; juvenile arthritis; GO KIDS; anti TNF alpha medications; juvenile psoriatic arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNTO 148 (Golimumab) (Experimental): All patients will receive golimumab 30 mg per square meter every 4 weeks from Week 0 through Week 12. Patients who have a clinical response at Week 16 and who are randomly allocated to golimumab, will receive 30 mg per square meter every 4 weeks through Week 48. Patients will continue to receive golimumab 30 mg per square meter after Week 48 in a long-term extension until Week 248. All patients will receive their fixed dose of commercial methotrexate throughout the study duration.
  Interventions: Drug: CNTO 148 (Golimumab); Drug: Methotrexate
- Placebo (Placebo Comparator): All patients will receive golimumab 30 mg per square meter every 4 weeks from Week 0 through Week 12. Patients who have a clinical response to golimumab at Week 16 and are randomly allocated to placebo, will receive placebo every 4 weeks through Week 48. However, patients receiving placebo and who will have lack/loss of clinical response will be eligible to receive golimumab 30 mg per square meter every 4 weeks through Week 48. At Week 48, patients do not have a clinical response will begin to receive golimumab 30 mg per square meter in a long-term extension until Week 248 and patients who have a clinical response will be discontinued from the study. All patients will receive their fixed dose of commercial methotrexate throughout the study duration.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: CNTO 148 (Golimumab) — Patients will receive subcutaneous (SC) (under the skin) injection of golimumab 30 mg per square meter every 4 weeks from Week 0 through Week 248.
  Arms: CNTO 148 (Golimumab)
Drug: Placebo — Patients who have a clinical response to golimumab at Week 16 and are randomly allocated to placebo, will receive SC injection of placebo every 4 weeks from Week 16 through Week 48.
  Arms: Placebo
Drug: Methotrexate — All patients will receive their fixed dose of commercial methotrexate (10 to 30 mg per square meter) weekly throughout the study duration.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of golimumab (CNTO 148) in patients who have active juvenile idiopathic arthritis (JIA) and at least 5 joints with active arthritis that have poor response to methotrexate.

DETAILED DESCRIPTION:
Approximately 170 juvenile patients will take part in the study worldwide. All patients will receive 30mg/m2 (milligrams per meter squared, up to 50 mg per dose) of golimumab subcutaneously (injection under the skin) every 4 weeks from Week 0 through Week 12. At Week 16, patients who have shown at least a 30 percent improvement in their signs and symptoms from when they started the study will be randomized to receive either placebo (sham medicine injection) or 30 mg/m2 of golimumab injections every 4 weeks from week 16 through week 48. If a patient gets markedly worse and is receiving placebo injections, they will be restarted on golimumab at the next scheduled visit and will continue on golimumab. Patients can leave the study at any time without question. Between the Week 48 analyses timepoint to Week 144, which is subsequently amended to Week 248, all patients will receive golimumab 30mg/meter squared, unless, by measurements, they have been nearly cured (clinical remission) by being on placebo, whereby they will be discontinued from the study. Patients may have a change in background treatment after Week 48 based on therapeutic effect. Patients will continue active treatment after Week 48 in a long-term extension until Week 144, which is subsequently amended to Week 248. All patients will receive their fixed dose of commercial methotrexate throughout the study duration. Safety will be monitored up to 152 week, which is subsequently amended to 256 weeks including drawing blood and looking at laboratory tests, vital signs (eg, blood pressure), and the frequency and type of adverse events (side effects).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis must have been before the patient's 16th birthday
* Disease duration of at least 6 months before study entry
* Must have 5 or more joints with active arthritis
* Must be taking a stable dose of methotrexate 10-30 mg/meter squared (patients with body surface area [BSA] 1.67 square meter or more must be taking a minimum of 15 mg/week of methotrexate)
* May take a stable dose of prednisone less than 10 mg/day 4 weeks prior to entry or may take a stable dose of NSAIDS (non-steroidal anti-inflammatory drugs) 2 weeks prior to entry
* Must have qualifying laboratory values at the first visit.

Exclusion Criteria:

* Have known allergies, hypersensitivity, or intolerance to golimumab or similar therapeutics
* Are pregnant or breast-feeding, or planning a pregnancy or fathering a child within 6 months after the last study agent administration
* Have initiated DMARDS and/or immunosuppressive therapy within 4 weeks prior to study initiation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 173 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (35):
- United States (7):
  - Los Angeles, California
  - San Francisco, California
  - Augusta, Georgia
  - Boston, Massachusetts
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
- Austria (2):
  - Bregenz
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Brazil (4):
  - Botucatu
  - Curitiba
  - Ribeirão Preto
  - Rio de Janeiro
- Canada (2):
  - Halifax, Nova Scotia
  - Toronto, Ontario
- Finland (2):
  - Helsinki
  - Oulu
- Germany (5):
  - Bad Bramstedt
  - Berlin
  - Bremen
  - Hamburg
  - Sankt Augustin
- Vilnius, Lithuania
- Mexico (3):
  - Mexico City
  - Monterrey
  - San Luis Potosí City
- Utrecht, Netherlands
- Poland (2):
  - Krakow
  - Lodz
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Samara

REFERENCES:
- [Derived] Brunner HI, Ruperto N, Tzaribachev N, Horneff G, Chasnyk VG, Panaviene V, Abud-Mendoza C, Reiff A, Alexeeva E, Rubio-Perez N, Keltsev V, Kingsbury DJ, Del Rocio Maldonado Velazquez M, Nikishina I, Silverman ED, Joos R, Smolewska E, Bandeira M, Minden K, van Royen-Kerkhof A, Emminger W, Foeldvari I, Lauwerys BR, Sztajnbok F, Gilmer KE, Xu Z, Leu JH, Kim L, Lamberth SL, Loza MJ, Lovell DJ, Martini A; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Subcutaneous golimumab for children with active polyarticular-course juvenile idiopathic arthritis: results of a multicentre, double-blind, randomised-withdrawal trial. Ann Rheum Dis. 2018 Jan;77(1):21-29. doi: 10.1136/annrheumdis-2016-210456. Epub 2017 May 15. PMID 28507219

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I: Participants Who Did Not Enter RW Period: Enrolled participants who did not enter randomized withdrawal (RW) period, including those who discontinued prior Week 16, and those who were non-responders (did not achieve an American College of Rheumatology [ACR] Ped 30 response) at Week 16.
- Group II: Placebo Subcutaneously (SC) + MTX: Participants who were treated with golimumab 30 milligram per square meter (mg/m^2) through Week 12 and were treated with placebo + Methotrexate (MTX) at Week 16 and continued on placebo + MTX through Week 48.
- Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX: Participants who were treated with golimumab 30 mg/m^2 through Week 12 and were treated with placebo + MTX at Week 16 and switched to golimumab 30 mg/m^2 + MTX at anytime during the study through Week 48. Adverse events are reported for participants who switched to golimumab 30 mg/m^2 + MTX at anytime during the study through Week 48.
- Group IV: Golimumab + MTX: Participants were treated with golimumab 30 mg/m^2 through Week 12 and who were treated with golimumab 30 mg/m^2 + MTX at Week 16 and continued on golimumab 30 mg/m^2 + MTX through Week 48.
Period: Overall Study
Arm/Group | Group I: Participants Who Did Not Enter RW Period | Group II: Placebo Subcutaneously (SC) + MTX | Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX | Group IV: Golimumab + MTX
Started | 19 | 11 | 65 | 78
Completed | 0 | 0 | 0 | 0
Not Completed | 19 | 11 | 65 | 78
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 2
Not completed — Lack of Efficacy | 14 | 1 | 2 | 3
Not completed — Adverse Event | 4 | 2 | 3 | 7
Not completed — Recovery | 0 | 6 | 0 | 0
Not completed — Study terminated by Sponsor | 0 | 2 | 56 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Participants Who Did Not Enter RW Period | Group II: Placebo Subcutaneously (SC) + MTX | Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX | Group IV: Golimumab + MTX | Total
Number analyzed (Participants) | 19 | 11 | 65 | 78 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (4.4) | 13.6 (2.2) | 10.7 (4.66) | 11.1 (4.43) | 11.2 (4.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 51 | 59 | 131
  Male | 4 | 5 | 14 | 19 | 42
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 0 | 2 | 2 | 5
  Belgium | 2 | 1 | 5 | 2 | 10
  Brazil | 1 | 0 | 3 | 4 | 8
  Canada | 2 | 0 | 0 | 5 | 7
  Finland | 0 | 0 | 0 | 1 | 1
  Germany | 4 | 7 | 14 | 24 | 49
  Lithuania | 0 | 0 | 6 | 4 | 10
  Mexico | 2 | 1 | 8 | 11 | 22
  Netherlands | 0 | 0 | 2 | 2 | 4
  Poland | 2 | 0 | 1 | 4 | 7
  Russian Federation | 4 | 1 | 12 | 12 | 29
  United States | 1 | 1 | 12 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 30 Response at Week 16 Who Did Not Experienced a Flare of Disease Through Week 48
Description: Percentage of participants with American College of Rheumatology (ACR) Ped 30 responders at Week 16 who did not experience a flare of disease between Week 16 and Week 48 calculated as number of participants with response and who did not experience flare divided by number of participants randomized. Flare of disease was defined as the worsening from Week 16 by 30% or more in 3 of the 6 ACR Pediatric (Ped) Core Set Variables with no more than 1 of the 6 ACR Ped Core Set variables improving by more than 30% at the time of the flare. The 6 variables are: physicians global assessment of disease, participants/parent global assessment of overall well-being, number of active joints (defined as either swelling, or in absence of swelling, limited range of motion associated with pain on motion or tenderness), number of joints with limited range of motion, physical function by childhood health assessment questionnaire, and erythrocyte sedimentation rate.
Time Frame: Week 16 through Week 48
Population: Intent-to-treat (ITT) population included all participants achieving American College of Rheumatology (ACR) Pediatric (Ped) 30 response who were randomized at Week 16.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received golimumab 30 mg per square meter every 4 weeks from Week 0 through Week 12. Participants who had a clinical response to golimumab at Week 16 and were randomly allocated to placebo, received placebo every 4 weeks through Week 48. However, participants receiving placebo and had flare received golimumab 30 mg/m^2 every 4 weeks through Week 48. At Week 48, participants who were receiving placebo not having a clinical remission switched to receive golimumab 30 mg/m^2 in a long-term extension until Week 248 and participants who were receiving placebo and had a clinical remission discontinued from the study. All participants received their fixed dose of commercial methotrexate throughout the study duration.
- CNTO 148 (Golimumab): Participants received golimumab 30 milligram per square meter (mg/m^2) every 4 weeks from Week 0 through Week 12. Participants who had a clinical response at Week 16 and who were randomly allocated to golimumab, received 30 mg/m^2 every 4 weeks through Week 48. Participants continued receiving golimumab 30 mg/m^2 after Week 48 in a long-term extension until Week 248. All participants received their fixed dose of commercial methotrexate throughout the study duration.
Arm/Group | Placebo | CNTO 148 (Golimumab)
Number analyzed (Participants) | 76 | 78
Percentage of Participants | 52.6 | 59.0

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 30 Response at Week 48
Description: Percentage of participants with ACR 30 response at Week 48 was calculated as number of participants with ACR 30 response at Week 48 divided by number of participants randomized. ACR Ped 30 response was defined as the worsening from Week 16 by 30% or more in 3 of the 6 ACR Pediatric (Ped) Core Set Variables with no more than 1 of the 6 ACR Ped Core Set variables improving by more than 30% at the time of the flare. The 6 variables are: physicians global assessment of disease, participants/parent global assessment of overall well-being, number of active joints (defined as either swelling, or in absence of swelling, limited range of motion associated with pain on motion or tenderness), number of joints with limited range of motion, physical function by childhood health assessment questionnaire, and erythrocyte sedimentation rate.
Time Frame: Week 16 through Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | CNTO 148 (Golimumab)
Number analyzed (Participants) | 76 | 78
Percentage of Participants | 55.3 | 52.6

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 30 Response Who Had Inactive Disease at Week 48
Description: Inactive disease is indicated by the presence of all of the following: no joints with active arthritis; no fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to juvenile idiopathic arthritis; no active uveitis (eye disease), normal erythrocyte sedimentation rate or C-reactive protein; physician global assessment of disease activity indicating no active disease; and duration of morning stiffness less than 15 minutes.
Time Frame: Week 16 through Week 48
Population: ITT population included all participants achieving ACR Ped 30 response who were randomized at Week 16.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | CNTO 148 (Golimumab)
Number analyzed (Participants) | 76 | 78
Percentage of Participants | 27.6 | 39.7

4. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission While on Medication for Juvenile Idiopathic Arthritis (JIA) at Week 48
Description: Clinical remission while on medication for JIA is defined as inactive disease at each visit for a period of 6 months or more while on medication. Inactive disease is indicated by the presence of all of the following: no joints with active arthritis; no fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to juvenile idiopathic arthritis; no active uveitis (eye disease), normal erythrocyte sedimentation rate or C-reactive protein; physician global assessment of disease activity indicating no active disease; and duration of morning stiffness less than 15 minutes.
Time Frame: Week 16 through Week 48
Population: ITT population included all participants achieving ACR Ped 30 response who were randomized at Week 16.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | CNTO 148 (Golimumab)
Number analyzed (Participants) | 76 | 78
Percentage of Participants | 11.8 | 12.8

ADVERSE EVENTS:
Time Frame: Day 1 up to Database lock [DBL] (approximately Week 184)
Description: Safety population included all participants who received at least one dose of either placebo or golimumab. One participant in the placebo + MTX group received golimumab 30 mg/m^2 + MTX and was included in group 3 in safety population.
Arm/Group | Group I: Participants Who Did Not Enter RW Period | Group II: Placebo Subcutaneously (SC) + MTX | Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX | Group IV: Golimumab + MTX
Serious Adverse Events (participants affected / at risk) | 4/19 | 2/10 | 15/66 | 18/78
Other Adverse Events (participants affected / at risk) | 14/19 | 9/10 | 60/66 | 68/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Participants Who Did Not Enter RW Period (N=19) | Group II: Placebo Subcutaneously (SC) + MTX (N=10) | Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX (N=66) | Group IV: Golimumab + MTX (N=78)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Gallbladder oedema (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6 | 8
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Somatoform disorder neurologic (Psychiatric disorders) | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Participants Who Did Not Enter RW Period (N=19) | Group II: Placebo Subcutaneously (SC) + MTX (N=10) | Group III: Placebo + MTX -> Golimumab 30 mg/m^2 + MTX (N=66) | Group IV: Golimumab + MTX (N=78)
Pharyngitis (Infections and infestations) | 0 | 0 | 6 | 9
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 9 | 10
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 4 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 4 | 10
Sinusitis (Infections and infestations) | 0 | 0 | 7 | 8
Tonsillitis (Infections and infestations) | 0 | 0 | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 25 | 20
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 4
Viral infection (Infections and infestations) | 0 | 0 | 4 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 7
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 3 | 6
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 11 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 6
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 10 | 15
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 3
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 5 | 7
Erythema of eyelid (Eye disorders) | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 10 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 5 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 9 | 7
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 7 | 11
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 13 | 12
Influenza like illness (General disorders) | 0 | 0 | 8 | 0
Injection site erythema (General disorders) | 1 | 0 | 1 | 2
Injection site reaction (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 15 | 9
Serositis (General disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1 | 3 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 4 | 6
Gastroenteritis (Infections and infestations) | 2 | 1 | 6 | 8
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 6 | 2
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 7
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 3 | 18 | 21
Otitis media (Infections and infestations) | 0 | 0 | 5 | 6
Paronychia (Infections and infestations) | 1 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less